CLINICAL TRIAL: NCT06882720
Title: Effects of Otago-based Multicomponent Exercise on Sarcopenia in Pre-Frailty Older Adults in Nursing Homes: A Randomized Controlled Trial
Acronym: PA&P-F&SP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Collaborators: Kunming Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AWFiS/2025_3_ZO
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-03

CONDITIONS: Pre-Frailty; Sarcopenia in Elderly
Keywords: Pre-Frailty; Sarcopenia; Multicomponent Exercise; Elderly People
MeSH Terms: conditions — Sarcopenia | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Otago-based Multicomponent Exercise (Experimental): The intervention is based on the Otago Exercise program, which includes cardiopulmonary exercises, resistance exercises, and balance training, with an additional eight resistance exercises.
  Interventions: Behavioral: Exercise
- Control group (No Intervention): Give only the physical activity necessary for daily living.

INTERVENTIONS:
Behavioral: Exercise — Cardiorespiratory exercises include walking at a normal pace for 30 minutes three times a week, or three 10-minute sessions. The resistance exercises involve five leg muscle strengthening exercises, including knee extensors, knee flexors, hip adductors, ankle plantar flexors, and ankle dorsolflexors, performed 8-10 times, 1-2 sets, 3 times a week, with 1 day intervals in between. Balance training includes 12 exercises such as kneeling, walking backwards, walking and turning, walking sideways, tandem standing (heel-toe standing), tandem walking (heel-toe walking), standing on one leg, walking on the heel, and walking on the tip of the foot. Only 1 set of 1 exercise, 3 times a week, 1 day interval in between. Add 4 upper body strength exercises and 4 lower body strength exercises to the OEP, using water bottles and elastic bands as AIDS. Each movement is completed 8-12 times, 1-3 sets, 3 times a week, 1 day apart.
  Arms: Otago-based Multicomponent Exercise

SUMMARY:
The objective of this clinical trial is to understand the efficacy of a targeted exercise program (Otago exercise program+Strength training) in elderly people with prefrailty and sarcopenia. The trial aims to answer the following main questions:

* Is OEP+ST effective in elderly people with prefrailty and sarcopenia?
* In what areas did participants improve during the OEP+ST intervention?

Researchers will randomly assign participants to an experimental group (OEP+ST) and a control group (daily care only) for comparison to see the effects of this intervention.

Participants in the EG group will:

* Exercise 3 times a week for 1 hour each time (including 10 minutes of warm-up, 40 minutes of exercise and 10 minutes of stretching) At the same time, it is necessary to walk for 30-40 minutes three times a week. It lasts for three months.
* Test and record their condition (including frailty, body composition, physical function, quality of life) before and after the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Participants were diagnosed with pre-existing frailty (Fried score 1-2); At the same time, they were also diagnosed with sarcopenia (according to AWGS Asian Sarcopenia Diagnostic Criteria 2019 edition: Grip strength: male < 28kg, female < 18kg; SMI: Male < 7.0kg/m2, female < 5.4kg/m2; Walking speed ≤1.0 m/s; 5 sit-up test times ≥12s); Simple mental status examination (MMSE score ≥21); There are no absolute contraindications to physical exercise (chest pain, chest tightness, palpitations, dyspnea, syncope, high fever, severe cough, severe diarrhea, gross hematuria, radiating pain in waist and legs, fracture, etc.).

Exclusion Criteria:

* Uncontrolled high blood pressure. Coronary artery disease. Rheumatoid arthritis. Type 2 diabetes. Respiratory diseases and lung diseases. Are taking or have used antibiotics and/or antifungal therapy in the past 4 weeks.

Unwillingness to stick to a prescribed schedule.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-28 (Actual)

PRIMARY OUTCOMES:
Gait Speed | From enrollment to the end of treatment at 2 weeks
  In order to harmonize the pace measurement method, the 2019 Asian Sarcopenia Working Group recommends the time it takes to walk 6 meters at a normal pace from moving as a measure of average pace. The test is carried out in an inspection room that is more than 8 meters long. Crutches that participants normally use can also be used. The start and end of the 6-meter distance are clearly marked. Subjects stand with their toes touching the starting line, and after being instructed to move forward at their usual speed, subjects start walking, inspectors start timing, and when subjects fully cross the 6-meter mark with one foot, inspectors stop timing. The test is performed twice, recording the shortest time (in seconds) required to complete each distance. The smaller the value, the faster the walking speed, the better the physical ability.
Skeletal muscle index | From enrollment to the end of treatment at 2 weeks
  The formula for calculating SMI in InBody is as follows: SMI= sum of segmental muscle mass (two arms and two legs) ÷ square of height.
Hand Strength | From enrollment to the end of treatment at 2 weeks
  HS was measured to estimate muscle strength and was performed with a hand dynamometer (Jamar Plus Digital Hand Dynamometer, Sammons Preston, USA). During the HS test, participants had to hold the dynamometer in their hand with the arm stretched parallel to the body while being instructed to stand upright. This measure was performed three times on the dominant hand with a rest interval of 1 min between measurements; finally, the best performance was used as the maximum peak (PK) of HS (in kg). The statistical analysis also included mean peak (mean PK).The higher the grip strength value, the greater the muscle strength, the better the physical ability.
Skeletal Muscle Mass | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 770 analyzer (InBody Co. Seoul, Korea), participants wore light clothing and no shoes.The higher the number, the more muscle the human body has.The ideal skeletal muscle content for men is 47% of standard body weight and 42% of standard body weight for women. A 10% move up or down is considered normal.

SECONDARY OUTCOMES:
Body Fat Mass | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 770 analyzer (InBody Co. Seoul, Korea), participants wore light clothing and no shoes.The higher the value of this index, the higher the body fat content.
Skeletal Lean Mass | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 770 analyzer (InBody Co. Seoul, Korea), participants wore light clothing and no shoes. The calculation method of SLM is different from that of SMM. The SLM in InBody report paper is the sum of protein, body water, and extracosseous inorganic salts. The ideal SLM for men is 80% of standard body weight and 72% of standard body weight for women. A 10% move up or down is considered normal.
Fat-Free Mass | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 770 analyzer (InBody Co. Seoul, Korea), participants wore light clothing and no shoes. The higher the value of this index, the heavier the body weight without fat.
TUG | From enrollment to the end of treatment at 2 weeks
  Time up and go.The TUG test measures the time(s) required for a subject to rise from a chair, walk 3 m, turn around, walk back to the chair, and sit down. It has been shown to be a predictor of sarcopenia in hospitalized patients with a mean age of 70.4±7.7 years.The smaller the value, the shorter the completion time, and the better the physical function.
ArmCurl | From enrollment to the end of treatment at 2 weeks
  Participants were asked to sit in a chair holding a 2KG weight with one arm and complete the maximum number of arm curls within 30 seconds. The greater the number of bends, the better the upper body strength may prove.
6MWT | From enrollment to the end of treatment at 2 weeks
  6MWT is used to assess an individual's cardiopulmonary function, exercise tolerance, and overall functional status. It measures the distance patients walk at maximum capacity in six minutes, reflecting their daily activity endurance and the adaptability of their cardiorespiratory system. For a round trip walk in a 50-meter long corridor, the recorder records the exact distance (meters) in 6 minutes. The reference value for healthy elderly people is 400-500 meters for men and 350-450 meters for women. The reference value for the elderly in the early stage of frailty is: men: 300-400 meters, women: 250-350 meters.
5 STS | From enrollment to the end of treatment at 2 weeks
  First sit in a chair of the appropriate height, complete 5 consecutive standing and sitting movements, and finally finish in a sitting position, during which no chair is allowed to be held by hand. Record how long it takes to complete the action. The completion time of Pre-Frailty Older Adults is ≥12-15 seconds, if it is greater than 15 seconds, it means that there is a risk of falling, and the risk of limited activity is higher.
TandemBalance | From enrollment to the end of treatment at 2 weeks
  Participants used the "toe" stick to the "heel" in a straight line walking way, with the fastest speed to complete 2 meters. The smaller the value, the faster the walking speed, which may represent better balance ability.

OTHER OUTCOMES:
Body Mass Index | From enrollment to the end of treatment at 2 weeks
  Using the Octupole Bioimpedance InBody 770 analyzer (InBody Co. Seoul, Korea), participants wore light clothing and no shoes. The average person's BMI is usually between 18 and 23.
EQ-5D-5L | From enrollment to the end of treatment at 2 weeks
  EQ-5D-5L is a quality of life scale that measures mobility, self-care, daily living, pain, anxiety and depression. A utility value of 0 (death) to 1 (full health) is converted into a health state through a "value set" developed by countries (some states may <0, indicating worse than death). The evaluation criteria of utility value adopted in this study are applicable to Asian population. The utility value of the elderly in the early stage of frailty ranges from 0.72 to 0.8, and the higher the number, the better the quality of life.
SPPB（Short Physical Performance Battery） | From enrollment to the end of treatment at 2 weeks
  SPPB Standardized tool for assessing lower limb function, balance, and mobility in older adults, developed by the National Institute on Aging. Based on a combined score of three simple tests, it can predict the risk of falls, disability, hospitalization and even death. It included a balance test, a 4-meter walking test, and a chair standing test five times. On a scale of 0-12, the lower the score, the worse the fitness. Older people in the early stages of frailty usually score 7-9.
Fried | From enrollment to the end of treatment at 2 weeks
  Fried Scale is a classic scale for evaluating the frailty of the elderly. It helps identify frailty of the elderly by measuring five physiological indicators (involuntary weight loss, weakened grip strength, fatigue, decreased walking speed, and decreased physical activity), so as to predict adverse health outcomes such as falls, disability, hospitalization and death. When each indicator reaches the specified threshold, 1 score is recorded. The higher the score, the more weak it is. 1-2 is classified as the Pre-frailty.

CONTACTS AND LOCATIONS:
Locations (1):
- Kunming Medical University, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No
This study involves the privacy of the participants and therefore cannot be shared.

REFERENCES:
- [Background] Saez de Asteasu ML, Martinez-Velilla N, Zambom-Ferraresi F, Garcia-Alonso Y, Galbete A, Ramirez-Velez R, Cadore EL, Izquierdo M. Short-Term Multicomponent Exercise Impact on Muscle Function and Structure in Hospitalized Older at Risk of Acute Sarcopenia. J Cachexia Sarcopenia Muscle. 2024 Dec;15(6):2586-2594. doi: 10.1002/jcsm.13602. Epub 2024 Oct 13. PMID 39400535
- [Background] Zou Z, Chen Z, Ni Z, Hou Y, Zhang Q. The effect of group-based Otago exercise program on fear of falling and physical function among older adults living in nursing homes: A pilot trial. Geriatr Nurs. 2022 Jan-Feb;43:288-292. doi: 10.1016/j.gerinurse.2021.12.011. Epub 2021 Dec 30. PMID 34974397